CLINICAL TRIAL: NCT03896503
Title: Randomized Phase II Trial of Topotecan Plus M6620 (VX-970, Berzosertib) Vs. Topotecan Alone in Patients With Relapsed Small-Cell Lung Cancer
Brief Title: Randomized Trial of Topotecan With M6620, an ATR Kinase Inhibitor, in Small Cell Lung Cancers and Small Cell Cancers Outside of the Lungs
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-01769; NCI-2019-01769 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-C-0009; 10268 (Other: National Cancer Institute LAO); 10268 (Other: CTEP); ZIABC011078 (NIH); NCT04162041 (obsolete NCT alias)
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Results first posted 2024-11-13 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-07

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma; Extrapulmonary Small Cell Neuroendocrine Carcinoma; Limited Stage Lung Small Cell Carcinoma; Platinum-Resistant Lung Small Cell Carcinoma; Platinum-Sensitive Lung Small Cell Carcinoma; Recurrent Lung Small Cell Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — berzosertib; Biopsy; Specimen Handling; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort I Arm I (topotecan hydrochloride) (Active Comparator): Participants receive topotecan hydrochloride IV over 30 minutes on days 1-5. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Participants may crossover to Arm II at disease progression. Participants undergo a CT scan during screening and on study as well as a tumor biopsy during screening. Participants may also undergo blood sample collection during screening and on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Topotecan Hydrochloride
- Cohort I Arm II (topotecan hydrochloride, berzosertib (M6620)) (Experimental): Participants receive topotecan hydrochloride IV over 30 minutes on days 1-5 and berzosertib (M6620) IV over 60 minutes on days 2 and 5. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Participants undergo a CT scan during screening and on study as well as a tumor biopsy during screening. Participants may also undergo blood sample collection during screening and on study.
  Interventions: Drug: Berzosertib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Topotecan Hydrochloride
- Cohort II (exploratory cohort: topotecan, berzosertib (M6620)) (Experimental): Cohort II: Participants receive topotecan hydrochloride IV over 30 minutes on days 1-5 and berzosertib (M6620) IV over 60 minutes on days 2 and 5. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Participants undergo a CT scan during screening and on study as well as a tumor biopsy during screening. Participants may also undergo blood sample collection during screening and on study.
  Interventions: Drug: Berzosertib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Topotecan Hydrochloride

INTERVENTIONS:
Drug: Berzosertib — Given IV
  Other Names: 2-Pyrazinamine, 3-(3-(4-((Methylamino)methyl)phenyl)-5-isoxazolyl)-5-(4-((1-methylethyl)sulfonyl)phenyl)-; M 6620; M6620; VX 970; VX-970; VX970
  Arms: Cohort I Arm II (topotecan hydrochloride, berzosertib (M6620)); Cohort II (exploratory cohort: topotecan, berzosertib (M6620))
Procedure: Biopsy Procedure — Undergo a tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo a CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Evotopin; Hycamptamine; Hycamtin; Nogitecan Hydrochloride; Potactasol; SKF S 104864 A; SKF S-104864-A; SKF S104864A; Topotec; Topotecan HCl; topotecan hydrochloride (oral)

SUMMARY:
This phase II trial studies how well berzosertib (M6620) works when given in combination with topotecan hydrochloride (topotecan) compared with topotecan alone in treating patients with small cell lung cancer that has come back (relapsed), or small cell cancer that arises from a site other than the lung (extrapulmonary). Drugs used in chemotherapy, such as topotecan hydrochloride, work by damaging the DNA (deoxyribonucleic acid) in tumor cells, causing those cells to die and the tumor to shrink. However, some tumor cells can become less affected by chemotherapy because they have ways to repair the damaged DNA. The addition of M6620 could help topotecan hydrochloride shrink the cancer and prevent it from returning by blocking enzymes needed for DNA repair.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the combination of berzosertib (M6620) with topotecan hydrochloride (topotecan) will result in an improvement in progression-free survival (PFS) compared to topotecan alone in patients with relapsed small cell lung cancer (SCLC).

SECONDARY OBJECTIVE:

I. To determine the objective response rate (ORR) and overall survival (OS) with the combination of M6220 and topotecan in patients with relapsed SCLC and extrapulmonary small cell cancers.

EXPLORATORY OBJECTIVES:

I. To perform molecular profiling assays on malignant and normal tissues, including, but not limited to ribonucleic acid (RNA) sequencing (RNA-Seq):

Ia. To assess expression of genes Schlafen family member 11 (SLFN11), MYC, and ataxia-telangiectasia mutated (ATM) among others.

Ib. To identify potential predictive biomarkers of response to a combination of M6620 with topotecan.

Ic. Identify mechanisms of drug sensitivity and resistance using deoxyribonucleic acid (DNA)- and RNA-based assessment platforms.

II. To contribute genetic analysis data from de-identified biospecimens to Genomic Data Commons (GDC), a well annotated cancer molecular and clinical data repository, for current and future research; specimens will be annotated with key clinical data, including presentation, diagnosis, staging, summary treatment, and if possible, outcome.

III. To bank formalin-fixed, paraffin-embedded (FFPE) tissue, blood (for cell-free DNA analysis), and nucleic acids obtained from patients at the Early-Phase and Experimental Clinical Trials (EET) Biobank at Nationwide Children's Hospital.

IV. To characterize circulating cell-free DNA (cfDNA) and circulating tumor cells in patients with relapsed SCLC and extrapulmonary small cell cancers.

V. To identify potential predictive biomarkers of response to a combination of M6620 with topotecan in patients with extrapulmonary small cell cancers.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients with SCLC are randomized to 1 of 2 arms.

ARM I: Participants receive topotecan hydrochloride intravenously (IV) over 30 minutes on days 1-5. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Participants may crossover to Arm II at disease progression. Participants undergo a computed tomography (CT) scan during screening and on study as well as a tumor biopsy during screening. Participants may also undergo blood sample collection during screening and on study.

ARM II: Participants receive topotecan hydrochloride IV over 30 minutes on days 1-5 and berzosertib (M6620) IV over 60 minutes on days 2 and 5. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Participants undergo a CT scan during screening and on study as well as a tumor biopsy during screening. Participants may also undergo blood sample collection during screening and on study.

COHORT II (Patients with extrapulmonary small cell cancer): Participants receive topotecan hydrochloride IV over 30 minutes on days 1-5 and berzosertib (M6620) IV over 60 minutes on days 2 and 5. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Participants undergo a CT scan during screening and on study as well as a tumor biopsy during screening. Participants may also undergo blood sample collection during screening and on study.

After completion of study treatment, patients are followed up at 4 weeks and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled to the primary cohort must have limited- or extensive-disease SCLC at diagnosis, with relapse at study entry with measurable disease at random assignment per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Both platinum-sensitive and platinum-resistant patients will be included
* Patients with extrapulmonary small cell cancers (cancers with small cell morphology and arising outside the lung, such as small cell prostate, bladder, etc.) will be eligible for the exploratory cohort
* Patients must be >= 18 years of age because no dosing or adverse event data are currently available on the use of M6620 in combination with topotecan in patients <18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Hemoglobin >= 9.0 g/dL - patients may receive transfusion to meet the hemoglobin (Hb) eligibility
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 2 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional upper limit of normal (ULN)
* Creatinine =< institutional ULN OR
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-positive subjects on combination antiretroviral therapy are eligible as long as they are on effective anti-retroviral therapy with undetectable viral load within 6 months and there is no drug-drug interaction with M6220
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* The effects of M6620 on the developing human fetus are unknown. For this reason and because DNA-damage response (DDR) inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months after completion of M6620 administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 6 months after completion of M6620 administration
* Patients with treated brain metastases are eligible if they are symptomatically stable while off steroid therapy for a minimum of 21 days
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with symptomatic brain metastasis are not eligible due to their extremely poor prognosis and since it is unclear whether the investigational agent penetrates the blood-brain barrier. However, subjects who have had treatment for their brain metastasis and are symptomatically stable while off steroid therapy for a minimum of 21 days may be enrolled
* Patients who have received prior topotecan therapy
* Patients who have had chemotherapy or radiotherapy within 3 weeks prior to enrollment.

  * Note: Patients who have had palliative radiotherapy may be included as long as they have recovered from any radiotherapy related adverse events (allow at least a week between radiotherapy completion and study treatment)
* Patients who have not recovered from adverse events due to prior anti-cancer therapy except hair loss and peripheral neuropathy (i.e., have residual toxicities > grade 1)
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to M6620 or topotecan used in study
* M6620 is primarily metabolized by cytochrome P450 3A4 (CYP3A4); therefore, concomitant administration with strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir) or inducers of CYP3A4 (e.g., rifampin, phenytoin, carbamazepine, phenobarbital, St. John's wort) should be avoided. Patients requiring any medications or substances that are strong inhibitors or inducers of CYP3A during the course of the study are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference for a list of drugs to avoid or of which to minimize use. The Patient Drug Interactions Handout and Wallet Card should be provided to patients. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness
* Pregnant women are excluded from this study because M6620 as a DDR inhibitor may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M6620, breastfeeding should be discontinued if the mother is treated with M6620. These potential risks may also apply to topotecan used in this study
* Patients with high grade neuroendocrine cancers, but with no small cell morphology will not be eligible
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Patients with Li-Fraumeni syndrome will not be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2026-06-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anish Thomas, Principal Investigator — National Cancer Institute LAO
Locations (33):
- United States (33):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - NCI - Center for Cancer Research, Bethesda, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Wake Forest Baptist Health - Hematology Oncology - Statesville, Statesville, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Takahashi N, Hao Z, Villaruz LC, Zhang J, Ruiz J, Petty WJ, Mamdani H, Riess JW, Nieva J, Pachecho JM, Fuld AD, Shum E, Chauhan A, Nichols S, Shimellis H, McGlone J, Sciuto L, Pinkiert D, Graham C, Shelat M, Kattappuram R, Abel M, Schroeder B, Upadhyay D, Krishnamurthy M, Sharma AK, Kumar R, Malin J, Schultz CW, Goyal S, Redon CE, Pommier Y, Aladjem MI, Gore SD, Steinberg SM, Vilimas R, Desai P, Thomas A. Berzosertib Plus Topotecan vs Topotecan Alone in Patients With Relapsed Small Cell Lung Cancer: A Randomized Clinical Trial. JAMA Oncol. 2023 Dec 1;9(12):1669-1677. doi: 10.1001/jamaoncol.2023.4025. PMID 37824137

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 104 participants were enrolled, and 82/104 participants were treated as shown in the Participant Flow table.
Groups:
- Platinum Response - Sensitive: Topotecan Monotherapy: Cohort I, Arm I (topotecan hydrochloride) Participants with pulmonary disease receive topotecan hydrochloride intravenously (IV) over 30 minutes on days 1-5. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Participants may crossover to Arm II at disease progression. Participants undergo a computed tomography (CT) scan during screening and on study as well as a tumor biopsy during screening. Participants may also undergo blood sample collection during screening and on study.
- Platinum Response - Sensitive: Topotecan & M6620 (VX-970) Combination Therapy: Cohort I, Arm II (topotecan hydrochloride & Berzosertib (M6620) Participants with pulmonary disease receive topotecan hydrochloride intravenously (IV) over 30 minutes on days 1-5 and Berzosertib (M6620) IV over 60 minutes on days 2 and 5. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Participants undergo a computed tomography (CT) scan during screening and on study as well as a tumor biopsy during screening. Participants may also undergo blood sample collection during screening and on study.
- Platinum Response - Sensitive: Enrolled But Not Treated; Platinum Response - Resistant: Enrolled But Not Treated: Participants with pulmonary disease were enrolled but not treated.
- Platinum Response - Resistant: Topotecan Monotherapy: Arm I (topotecan hydrochloride) Participants with pulmonary disease receive topotecan hydrochloride intravenously (IV) over 30 minutes on days 1-5. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Participants may crossover to Arm II at disease progression. Participants undergo a computed tomography (CT) scan during screening and on study as well as a tumor biopsy during screening. Participants may also undergo blood sample collection during screening and on study.
- Platinum Response - Resistant: Topotecan & M6620 (VX-970) Combination Therapy: Arm II (topotecan hydrochloride & Berzosertib (M6620) Participants with pulmonary disease receive topotecan hydrochloride intravenously (IV) over 30 minutes on days 1-5 and Berzosertib (M6620) IV over 60 minutes on days 2 and 5. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Participants undergo a computed tomography (CT) scan during screening and on study as well as a tumor biopsy during screening. Participants may also undergo blood sample collection during screening and on study.
- Exploratory Cohort: Topotecan & M6620 (VX-970) Combination Therapy: Arm II (topotecan hydrochloride & Berzosertib (M6620) Participants receive topotecan hydrochloride intravenously (IV) over 30 minutes on days 1-5 and Berzosertib (M6620) IV over 60 minutes on days 2 and 5. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Participants undergo a computed tomography (CT) scan during screening and on study as well as a tumor biopsy during screening. Participants may also undergo blood sample collection during screening and on study.
- Exploratory Cohort: Enrolled But Not Treated: Participants were enrolled but not treated.
Period: Initial Subgroup and Arm Enrollment
Arm/Group | Platinum Response - Sensitive: Topotecan Monotherapy | Platinum Response - Sensitive: Topotecan & M6620 (VX-970) Combination Therapy | Platinum Response - Sensitive: Enrolled But Not Treated | Platinum Response - Resistant: Topotecan Monotherapy | Platinum Response - Resistant: Topotecan & M6620 (VX-970) Combination Therapy | Platinum Response - Resistant: Enrolled But Not Treated | Exploratory Cohort: Topotecan & M6620 (VX-970) Combination Therapy | Exploratory Cohort: Enrolled But Not Treated
Started | 10 | 20 | 10 | 11 | 23 | 9 | 18 | 3
Not Treated | 1 | 0 | 10 | 1 | 2 | 9 | 2 | 3
Off Treatment | 7 | 17 | 0 | 10 | 0 | 0 | 16 | 0
Completed | 7 | 18 | 0 | 10 | 20 | 0 | 16 | 0
Not Completed | 3 | 2 | 10 | 1 | 3 | 9 | 2 | 3
Not completed — Disease progression before treatment | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — No treatment per protocol | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Late determination of ineligibility | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Declined to participate | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Not treated; participate found ineligible | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0
Not completed — Not treated; screen failure | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 2
Not completed — Refused further treatment | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Off treatment? other reasons withdrew consent | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not treated; death before treatment | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Not treated; participate found ineligible | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Off treatment; screen failure | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Period: Crossover Participants
Arm/Group | Platinum Response - Sensitive: Topotecan Monotherapy | Platinum Response - Sensitive: Topotecan & M6620 (VX-970) Combination Therapy | Platinum Response - Sensitive: Enrolled But Not Treated | Platinum Response - Resistant: Topotecan Monotherapy | Platinum Response - Resistant: Topotecan & M6620 (VX-970) Combination Therapy | Platinum Response - Resistant: Enrolled But Not Treated | Exploratory Cohort: Topotecan & M6620 (VX-970) Combination Therapy | Exploratory Cohort: Enrolled But Not Treated
Started | 0 | 5 | 0 | 0 | 6 | 0 | 0 | 0
Not Treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Off Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 5 | 0 | 0 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data was collected and is reported here for participants enrolled but not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Platinum Response - Sensitive: Topotecan Monotherapy | Platinum Response - Sensitive: Topotecan & M6620 (VX-970) Combination Therapy | Platinum Response - Sensitive: Enrolled But Not Treated | Platinum Response - Resistant: Topotecan Monotherapy | Platinum Response - Resistant: Topotecan & M6620 (VX-970) Combination Therapy | Platinum Response - Resistant: Enrolled But Not Treated | Exploratory Cohort: Topotecan & M6620 (VX-970) Combination Therapy | Exploratory Cohort: Enrolled But Not Treated | Total
Number analyzed (Participants) | 10 | 20 | 10 | 11 | 23 | 9 | 18 | 3 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 12 | 6 | 7 | 15 | 6 | 11 | 1 | 65
  >=65 years | 3 | 8 | 4 | 4 | 8 | 3 | 7 | 2 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (9.53) | 61.65 (9.05) | 63 (8.17) | 61.72 (7.00) | 60.60 (7.57) | 58.33 (8.83) | 57.94 (13.24) | 64.33 (2.49) | 60.16 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 5 | 5 | 10 | 3 | 5 | 0 | 41
  Male | 4 | 13 | 5 | 6 | 13 | 6 | 13 | 3 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 20 | 10 | 11 | 22 | 9 | 18 | 3 | 103
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 4 | 0 | 0 | 1 | 1 | 2 | 2 | 10
  White | 10 | 15 | 10 | 11 | 20 | 7 | 14 | 1 | 88
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 10 | 20 | 10 | 11 | 23 | 9 | 18 | 3 | 104

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Reported With 80% Confidence Interval
Description: The combination of M6620 with topotecan will be compared to topotecan alone in participants with relapsed small cell lung cancer (SCLC). Kaplan-Meier curves and a one-tailed log-rank test will be the primary analysis methods. PFS is defined as the duration of time from start of treatment to time of progression or death. whichever occurs first. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) and is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, and/or the appearance of one or more new lesions.
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed at 6 months after last participant has enrolled; up to 2 years for pulmonary cohort and up 31.5 months for Exploratory Cohort.
Population: Participants enrolled but not treated are not reported for this outcome measure. Six participants from the groups reported below were not evaluable for this outcome measure. Participants who have results reported were placed into categories per initial randomization. Exploratory cohort consists of participants with extrapulmonary disease and were not randomized to treatment.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Platinum Response - Sensitive: Topotecan Monotherapy | Platinum Response - Sensitive: Topotecan & M6620 (VX-970) Combination Therapy | Platinum Response - Resistant: Topotecan Monotherapy | Platinum Response - Resistant: Topotecan & M6620 (VX-970) Combination Therapy | Exploratory Cohort: Topotecan & M6620 (VX-970) Combination Therapy
Number analyzed (Participants) | 9 | 20 | 11 | 20 | 16
Months | 5.5 [2.6 to 6.0] | 4.4 [3.4 to 5.5] | 2.1 [1.3 to 3.0] | 2.7 [2.0 to 4.0] | 1.5 [1.4 to 1.8]

2. Primary Outcome: Progression-free Survival (PFS) Reported With 95% Confidence Interval
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Platinum Response - Sensitive: Topotecan Monotherapy | Platinum Response - Sensitive: Topotecan & M6620 (VX-970) Combination Therapy | Platinum Response - Resistant: Topotecan Monotherapy | Platinum Response - Resistant: Topotecan & M6620 (VX-970) Combination Therapy | Exploratory Cohort: Topotecan & M6620 (VX-970) Combination Therapy
Number analyzed (Participants) | 9 | 20 | 11 | 20 | 16
Months | 5.5 [1.2 to 9.6] | 4.4 [3.0 to 8.2] | 2.1 [0.9 to 4.1] | 2.7 [1.5 to 5.4] | 1.5 [1.3 to 2.9]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as percentage of participants who achieved either complete response (CR) or partial response (PR) as best response assessed using the revised Response Evaluation Criteria in Solid Tumors guideline (v 1.1). ORR percentage is calculated as the sum of the PR and CR rates, divided by the total number of participants who are evaluable for a response, multiplied by 100%. All participants included in the study must be assessed for response to treatment, even if there are major protocol treatment deviations or if they are ineligible. Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the diameters of target lesions. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive disease is at least a 20% increase in the sum of the diameters of target lesions.
Time Frame: Up to 2 years
Population: Participants enrolled but not treated are not reported for this outcome measure. Ten participants from the groups reported below were not evaluable for this outcome measure. Participants who have results reported were placed into categories per initial randomization. Exploratory cohort consists of participants with extrapulmonary disease and were not randomized to treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Platinum Response - Sensitive: Topotecan Monotherapy | Platinum Response - Sensitive: Topotecan & M6620 (VX-970) Combination Therapy | Platinum Response - Resistant: Topotecan Monotherapy | Platinum Response - Resistant: Topotecan & M6620 (VX-970) Combination Therapy | Exploratory Cohort: Topotecan & M6620 (VX-970) Combination Therapy
Number analyzed (Participants) | 8 | 20 | 10 | 19 | 15
Percentage of participants
  Complete Response | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Partial Response | 12.5 [0.3 to 52.7] | 35.0 [15.4 to 59.2] | 0 [0 to 30.9] | 15.8 [3.3 to 39.6] | 23.3 [1.7 to 40.5]

4. Secondary Outcome: Overall Survival (OS) Reported With 80% Confidence Interval
Description: OS is defined as time from randomization to death, regardless of cause.
Time Frame: Up to 2 years for pulmonary cohort and up 31.5 for Exploratory Cohort.
Population: as for outcome 1
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Platinum Response - Sensitive: Topotecan Monotherapy | Platinum Response - Sensitive: Topotecan & M6620 (VX-970) Combination Therapy | Platinum Response - Resistant: Topotecan Monotherapy | Platinum Response - Resistant: Topotecan & M6620 (VX-970) Combination Therapy | Exploratory Cohort: Topotecan & M6620 (VX-970) Combination Therapy
Number analyzed (Participants) | 9 | 20 | 11 | 20 | 16
Months | 6.5 [3.2 to 7.1] | 9.6 [8.0 to 11.4] | 4.6 [2.7 to 6.0] | 6.1 [3.7 to 11.8] | 6.7 [2.4 to 8.1]

5. Secondary Outcome: Overall Survival (OS) Reported With 95% Confidence Interval
Description: OS is defined as time from randomization to death, regardless of cause.
Time Frame: Up to 2 years for pulmonary cohort and up 31.5 for Exploratory Cohort
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Platinum Response - Sensitive: Topotecan Monotherapy | Platinum Response - Sensitive: Topotecan & M6620 (VX-970) Combination Therapy | Platinum Response - Resistant: Topotecan Monotherapy | Platinum Response - Resistant: Topotecan & M6620 (VX-970) Combination Therapy | Exploratory Cohort: Topotecan & M6620 (VX-970) Combination Therapy
Number analyzed (Participants) | 9 | 20 | 11 | 20 | 16
Months | 6.5 [1.2 to 9.6] | 9.6 [5.5 to 11.8] | 4.6 [1.4 to 6.2] | 6.1 [2.3 to 12.1] | 6.7 [2.2 to 9.4]

6. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, an average of 801.3 days.
Population: Participants enrolled but not treated are not reported for this outcome measure. Adverse events would not be monitored/assessed if the participant never received drug. Six participants (i.e., enrolled but not treated) from the groups reported below were not evaluable for this outcome measure. Participants who have results reported were placed into categories per initial randomization. Exploratory cohort consists of participants with extrapulmonary disease and were not randomized to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum Response - Sensitive: Topotecan Monotherapy | Platinum Response - Sensitive: Topotecan & M6620 (VX-970) Combination Therapy | Platinum Response - Resistant: Topotecan Monotherapy | Platinum Response - Resistant: Topotecan & M6620 (VX-970) Combination Therapy | Exploratory Cohort: Topotecan & M6620 (VX-970) Combination Therapy
Number analyzed (Participants) | 9 | 20 | 11 | 20 | 16
Participants | 8 | 20 | 11 | 19 | 16

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, an average of 801.3 days.
Description: Adverse events would not be monitored/assessed if the participant never received drug (i.e., enrolled but not treated). This is not a cross over study, rather there is an option to cross over, and exploratory data collected. 11 participants crossed over. Adverse events for cross over participants are represented in initial arm, and separately in the table below.
Groups:
- Platinum Response - Sensitive: Topotecan & M6620 Combination Therapy -Cross-over From Cohort 1 Arm I: Platinum Response - Sensitive: Topotecan & M6620 (VX-970) Combination Therapy -- Cross-over from Cohort 1 Arm I
- Platinum Response -Resistant: Topotecan & M6620 Combination Therapy - Cross-over From Cohort 2 Arm 1: Platinum Response - Resistant: Topotecan & M6620 (VX-970) Combination Therapy -- Cross-over from Cohort 2 Arm 1
Arm/Group | Platinum Response - Sensitive: Topotecan Monotherapy | Platinum Response - Sensitive: Topotecan & M6620 (VX-970) Combination Therapy | Platinum Response - Resistant: Topotecan Monotherapy | Platinum Response - Resistant: Topotecan & M6620 (VX-970) Combination Therapy | Exploratory Cohort: Topotecan & M6620 (VX-970) Combination Therapy | Platinum Response - Sensitive: Topotecan & M6620 Combination Therapy -Cross-over From Cohort 1 Arm I | Platinum Response -Resistant: Topotecan & M6620 Combination Therapy - Cross-over From Cohort 2 Arm 1
All-Cause Mortality (participants affected / at risk) | 9/9 | 19/20 | 11/11 | 19/20 | 15/16 | 5/5 | 6/6
Serious Adverse Events (participants affected / at risk) | 6/9 | 12/20 | 9/11 | 11/20 | 9/16 | 4/5 | 4/6
Other Adverse Events (participants affected / at risk) | 8/9 | 20/20 | 11/11 | 19/20 | 16/16 | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platinum Response - Sensitive: Topotecan Monotherapy (N=9) | Platinum Response - Sensitive: Topotecan & M6620 (VX-970) Combination Therapy (N=20) | Platinum Response - Resistant: Topotecan Monotherapy (N=11) | Platinum Response - Resistant: Topotecan & M6620 (VX-970) Combination Therapy (N=20) | Exploratory Cohort: Topotecan & M6620 (VX-970) Combination Therapy (N=16) | Platinum Response - Sensitive: Topotecan & M6620 Combination Therapy -Cross-over From Cohort 1 Arm I (N=5) | Platinum Response -Resistant: Topotecan & M6620 Combination Therapy - Cross-over From Cohort 2 Arm 1 (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 3 (4) | 4 (5) | 2 (2) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other, Increased Lactic Acid (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 5 (5) | 1 (1) | 3 (4) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mobitz type I (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Brain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 1 (2) | 3 (5) | 4 (5) | 2 (2) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stroke (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Thromboembolic event (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platinum Response - Sensitive: Topotecan Monotherapy (N=9) | Platinum Response - Sensitive: Topotecan & M6620 (VX-970) Combination Therapy (N=20) | Platinum Response - Resistant: Topotecan Monotherapy (N=11) | Platinum Response - Resistant: Topotecan & M6620 (VX-970) Combination Therapy (N=20) | Exploratory Cohort: Topotecan & M6620 (VX-970) Combination Therapy (N=16) | Platinum Response - Sensitive: Topotecan & M6620 Combination Therapy -Cross-over From Cohort 1 Arm I (N=5) | Platinum Response -Resistant: Topotecan & M6620 Combination Therapy - Cross-over From Cohort 2 Arm 1 (N=6)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 5 (9) | 3 (3) | 0 (0) | 7 (11) | 1 (1) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (10) | 6 (10) | 6 (8) | 3 (4) | 5 (6) | 1 (8) | 3 (3)
Alkaline phosphatase increased (Investigations) | 6 (13) | 10 (15) | 6 (8) | 3 (5) | 3 (5) | 4 (10) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 2 (2) | 4 (6) | 2 (3) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 8 (42) | 18 (80) | 9 (38) | 16 (81) | 12 (28) | 5 (33) | 5 (22)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 7 (9) | 3 (3) | 4 (4) | 4 (6) | 1 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (12) | 4 (5) | 3 (5) | 2 (4) | 3 (3) | 2 (7) | 2 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 6 (6) | 3 (4) | 7 (10) | 0 (0) | 3 (3)
Belching (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1) | 2 (5) | 2 (2) | 2 (2) | 0 (0) | 2 (5)
Blood bilirubin increased (Investigations) | 2 (5) | 2 (5) | 2 (11) | 2 (2) | 1 (4) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin T increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Chills (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 4 (5) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (6) | 8 (12) | 1 (1) | 2 (2) | 3 (6) | 3 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 3 (4) | 3 (4) | 3 (3) | 2 (2) | 2 (3)
Creatinine increased (Investigations) | 1 (1) | 3 (8) | 2 (3) | 1 (1) | 5 (8) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 5 (6) | 5 (6) | 4 (11) | 4 (8) | 1 (2) | 2 (2)
Dizziness (Nervous system disorders) | 1 (2) | 5 (6) | 4 (6) | 4 (6) | 3 (3) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 3 (4) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 5 (5) | 5 (7) | 5 (5) | 4 (8) | 3 (5) | 4 (6)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 4 (6) | 1 (1) | 4 (7) | 3 (4) | 1 (2) | 3 (5) | 2 (4)
Electrocardiogram T wave abnormal (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (4) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, R Eye Issue (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 1 (2) | 2 (5) | 0 (0) | 1 (1) | 1 (2)
Fatigue (General disorders) | 4 (4) | 13 (24) | 9 (20) | 11 (18) | 10 (15) | 2 (2) | 4 (9)
Fever (General disorders) | 1 (3) | 3 (4) | 2 (3) | 4 (6) | 3 (4) | 1 (3) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Cold sores on tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, Aches (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, Specify (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Burning and/or frequency with urination
General disorders and administration site conditions - Other, Specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Weak and shaky due to upset stomach and nausea
General disorders and administration site conditions - Other, catheter occulsion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3) | 1 (1) | 3 (4) | 4 (5) | 1 (1) | 1 (1)
Glucosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 7 (7) | 3 (4) | 4 (4) | 2 (5) | 1 (1) | 1 (1)
Heart failure (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4) | 6 (10) | 1 (2) | 3 (4) | 5 (6) | 1 (3) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 3 (6) | 2 (5) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 4 (5) | 2 (2) | 4 (4) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 2 (4) | 4 (6) | 1 (2) | 2 (10) | 3 (5) | 2 (4) | 1 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (11) | 5 (10) | 5 (10) | 4 (5) | 4 (12) | 3 (9) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (10) | 6 (16) | 7 (14) | 4 (6) | 6 (12) | 2 (7) | 4 (10)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 5 (15) | 4 (7) | 6 (13) | 7 (11) | 3 (4) | 3 (13) | 2 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (4) | 7 (17) | 4 (6) | 5 (7) | 2 (2) | 2 (4) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (11) | 9 (36) | 6 (10) | 7 (16) | 7 (9) | 2 (10) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (4) | 4 (5) | 2 (2) | 3 (3) | 5 (8) | 3 (4) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 7 (10) | 1 (1) | 4 (5) | 2 (2) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
INR increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 3 (4) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Investigations - Other, CK elevated (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, Increased ANC (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Investigations - Other, Increased PT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Investigations - Other, Increased WBC (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, LDH elevate (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, d.bili increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, lightheadedness (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 5 (11) | 1 (2) | 5 (12) | 1 (1) | 0 (0) | 1 (2)
Lipase increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 5 (25) | 15 (41) | 8 (33) | 11 (25) | 10 (22) | 3 (19) | 3 (16)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, Lactic Acid (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (7) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, RT shoulder stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 4 (7) | 9 (18) | 6 (6) | 10 (16) | 6 (10) | 3 (5) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (2) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Level IV left neck lymph node
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, numbness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, aphasia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (8) | 10 (16) | 6 (12) | 11 (15) | 9 (12) | 3 (5) | 3 (6)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (6) | 2 (3) | 3 (3) | 1 (1) | 1 (2) | 2 (3)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0
Otitis externa (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (7) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 3 (6) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Platelet count decreased (Investigations) | 7 (35) | 20 (71) | 11 (37) | 16 (67) | 14 (37) | 4 (29) | 6 (17)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, Catheter occlusion (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, Difficulty urinating (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, decreased urine output (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Complete post obstructive consolidation of right lower lobe
Respiratory, thoracic and mediastinal disorders - Other, Intermittent warm sensation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Pulmonary vascular congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, chest-shortness of breath w/exertion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (5) | 2 (2) | 1 (2) | 2 (2) | 3 (5) | 2 (5) | 1 (2)
Skin and subcutaneous tissue disorders - Other, Bee Stings (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Cellulitis-Rt Eyebrow (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Dermatitis rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Rash NOS on bilateral arms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Rash NOS on lower back (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Scalp Sensitivty (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Skin Lesions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, candidal intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, jaundice (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, port scab (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, sunburn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, suprapubic erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders - Other, pulmonary embolus (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 5 (6) | 3 (3) | 6 (13) | 2 (2) | 1 (2) | 2 (2)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (1) | 4 (7) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 6 (14) | 14 (28) | 7 (26) | 12 (22) | 11 (22) | 3 (9) | 4 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT03896503/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT03896503/ICF_002.pdf